CLINICAL TRIAL: NCT05551299
Title: Cholangiocarcinoma Treatment with Radiofrequency Ablation or Photodynamic Therapy: a Randomized Controlled Trial
Brief Title: Treatment of Non-resectable Bile Duct Cancer with Radiofrequency Ablation or Photodynamic Therapy
Acronym: CARP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Zentrum für Klinische Studien Leipzig (Other)
Responsible Party: Principal Investigator, Albrecht Hoffmeister, Prof. Dr. med., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARP; 2022-500107-50-00 (Other: EU CT Number (EMA)); 434336116 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft (DFG))
Record Dates: First submitted 2022-09-08; First posted 2022-09-22 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hilar Cholangiocarcinoma
Keywords: Hilar Cholangiocarcinoma; Radiofrequency ablation (RFA); Photodynamic therapy (PDT); Photosensitizer; Klatskin Tumor; Bile Duct Cancer
MeSH Terms: conditions — Klatskin Tumor; Bile Duct Neoplasms | interventions — Photosensitizing Agents; Photochemotherapy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photodynamic therapy (PDT) (Experimental): The index procedure in all patients at baseline includes stenting, using an endoscopic retrograde cholangio-pancreatography (ERCP) procedure. The Intervention is at least one PDT at baseline according to the clinical routine of the trial site.
  Interventions: Drug: Photosensitizer
- Radiofrequency ablation (RFA) (Experimental): The index procedure in all patients at baseline includes stenting, using an endoscopic retrograde cholangio-pancreatography (ERCP) procedure. The Intervention is at least one RFA at baseline according to the clinical routine of the trial site.
  Interventions: Procedure: Radiofrequency ablation (RFA)

INTERVENTIONS:
Drug: Photosensitizer — A photosensitizer, which is absorbed preferentially by tumour cells, is administered 24 - 48 hours prior to PDT. Light of a particular wavelength is then applied during endoscopic retrograde cholangiopancreatography (ERCP) to kill primarily cancer cells locally within the stenosis. Immediately after PDT treatment, new stents are inserted into all treated segments if needed.
  Other Names: Photodynamic therapy (PDT)
  Arms: Photodynamic therapy (PDT)
Procedure: Radiofrequency ablation (RFA) — RFA is also carried out as part of an ERCP. The RFA-probe is placed within the tumour stenosis and electrical current is applied. New stents are inserted into all treated segments if needed.
  Arms: Radiofrequency ablation (RFA)

SUMMARY:
Bile duct cancer is often diagnosed after curative options are no longer available. Stent therapy is used to keep the ducts open and can be combined with photodynamic therapy (PDT) to extend life expectancy. PDT requires an injection of photosensitizer after which light of a particular wavelength is applied endoscopically to kill the cancer cells. Drawbacks include not only high costs and poor availability, but foremost that patients have to avoid direct sunlight for a period of weeks. Radio frequency ablation (RFA) together with stent implantation constitutes an alternative by which the cancer cells are killed through heat, also applied endoscopically. The RFA technology is more widely available and easier to deploy. However, it has not been studied extensively and no randomized trials exist comparing the two methods. This trial will compare survival in patients with a particular bile duct cancer depending on whether they receive PDT or RFA. Moreover, data will be collected on side-effects and quality of life.

DETAILED DESCRIPTION:
Klatskin tumours are a form of bile duct cancer. They are generally not diagnosed until quite late and a curative operation is rarely a possibility. Their anatomic location usually results in bile duct obstruction and the aim of therapy is thus to keep the ducts open. This is accomplished through endoscopic retrograde cholangiopancreatography (ERCP) by implanting stents. Stent therapy combined with photodynamic therapy (PDT) extends life expectancy. PDT requires an injection of photosensitizer that is absorbed primarily by the cancer cells. Light of a particular wavelength is then applied with ERCP to kill the cancer cells. Drawbacks include not only high costs and poor availability, but foremost that patients have to avoid direct sunlight for a period of weeks. Radio frequency ablation (RFA) together with stent implantation constitutes an alternative by which the cancer cells are killed through heat applied during ERCP. The RFA technology is more widely available and easier to deploy. However, it has not been studied extensively and no randomized trials exist comparing the two methods. This trial will compare survival in patients with Klatskin tumours depending on whether they receive PDT or RFA. Moreover, data will be collected on side-effects and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Hilar cholangiocarcinoma (cytological or histological confirmation)
2. Surgery is not planned
3. Age ≥ 18 years
4. Written informed consent

Exclusion Criteria:

1. Tumour not accessible endoscopically
2. Known hypersensitivity to porphyrins or to any of the other ingredients of the photosensitizer chosen
3. Leukopenia (< 2000/mm3)
4. Thrombocytopenia (< 100,000 / mm³)
5. Severe, uncorrected coagulopathy (at the discretion of the physician)
6. Suspected erosion of major blood vessels, because of the risk of life-threatening mass haemorrhage exists
7. Porphyria (clinician's assessment) or other light-exacerbated diseases
8. Severely impaired liver and or kidney function (at the discretion of the physician)
9. Bedridden for more than 50% of the time (similar to ECOG (Eastern Cooperative Oncology Group) grade 3)
10. Planned surgical procedure within the next 30 days
11. Concurrent eye disease that will require a slit lamp examination within the next 30 days
12. Prior radiotherapy within the last four weeks
13. Previous PDT or RFA
14. Planned liver transplantation
15. Fertile women (within two years of their last menstruation) without appropriate contraceptive measures (implanon, injections, oral contraceptives, intrauterine devices, partner with vasectomy) while participating in the trial (participants using a hormone-based method have to be informed of possible effects of the trial medication on contraception)
16. Participation in other interventional trials
17. Patients under legal supervision or guardianship
18. Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | through study completion, an average of 1 year
  Hazard ratio from a Cox regression model will be used to compare randomization arms. Covariates will be stratification variables, classification of local inoperability, use of prophylactic antibiotics, Bismuth type and time between diagnosis and beginning RFA/PDT.

SECONDARY OUTCOMES:
Overall survival (complementary perspective: median survival time) | through study completion, an average of 1 year
  Estimates of the difference in median survival time between the groups will be based on the method of Chen and Zhang (PMID: 26983640).
Overall survival (complementary perspective: two-year overall survival) | up to two years
  Kaplan-Meier estimates will be used.
Overall survival (complementary perspective: restricted mean survival on a time horizon of two-years) | through study completion, an average of 1 year
  Kaplan-Meier estimates will be used (see e.g. PMID: 15690989)
Days alive and out of hospital up to two years | up to two years
  This constitutes a basic and easy to understand measure of quality of life. Only in-hospital stays will be included in this endpoint and the day of arrival and dismissal will each be counted. The source of data will be the hospital records, epicrisis and patient disclosure.
Quality of Life (QoL) measured using QLQ-C30 at various points in time after randomization (V2 (14 days), V3 (ca. 3 months), as a function of time after 6 months, adjusting for the baseline value) | through study completion, an average of 1 year
  Prolonging life is especially worthwhile if QoL is sufficiently good. The established cancer-specific Core Quality of Life questionnaire QLQ-C30 from the EORTC (European Organisation for Research will be used. Shortly after the index therapy (V2, V3), the difference between arms will be assessed. The requirement to stay indoors may affect QoL. At later points in time, a description per arm is of interest and will be based on a weighted mean of all available questionnaires, weighting according to calendar time.
Quality of Life (QoL) measured using FACT-Hep at various points in time after randomization (V2 (14 days), V3 (ca. 3 months), as a function of time after 6 months, adjusting for the baseline value) | through study completion, an average of 1 year
  Prolonging life is especially worthwhile if QoL is sufficiently good. The Functional Assessment of Cancer Therapy - Hepatobiliary (FACT-Hep) questionnaire, containing the hepatobiliary-specific cancer subscale, will be used as a second instrument for assessing QoL. Shortly after the index therapy (V2, V3), the difference between arms will be assessed. The requirement to stay indoors may affect QoL. At later points in time, a description per arm is of interest and will be based on a weighted mean of all available questionnaires, weighting according to calendar time.
Quality-adjusted life years (QALYs) | through study completion, an average of 1 year
  Using QALYs, a weighted measure of survival will be compared between RFA and PDT that takes QoL into account. The details will be provided in a Statistical Analysis Plan.
Stent patency based on clinician's assessment (e.g. cholangitis, cholestasis, ultrasound) | through study completion, an average of 1 year
  Stent patency provides one measure of the burden of the disease and efficacy of the treatment. Mean time to stent closure/replacement/death after last stent replacement will be analysed.
Laboratory parameter (leucocytes) | through study completion, an average of 1 year
  Changes in laboratory parameters after index treatment (V3) and as a function of time will be analysed and compared between randomization arms.
Laboratory parameter (haematocrit) | through study completion, an average of 1 year
  Changes in laboratory parameters after index treatment (V3) and as a function of time will be analysed and compared between randomization arms.
Laboratory parameter (haemoglobin) | through study completion, an average of 1 year
  Changes in laboratory parameters after index treatment (V3) and as a function of time will be analysed and compared between randomization arms.
Laboratory parameter (bilirubin) | through study completion, an average of 1 year
  Changes in laboratory parameters after index treatment (V3) and as a function of time will be analysed and compared between randomization arms.
Laboratory parameter (albumin) | through study completion, an average of 1 year
  Changes in laboratory parameters after index treatment (V3) and as a function of time will be analysed and compared between randomization arms.
Laboratory parameter (CA 19-9) | through study completion, an average of 1 year
  Changes in laboratory parameters after index treatment (V3) and as a function of time will be analysed and compared between randomization arms.
Laboratory parameter (CRP) | through study completion, an average of 1 year
  Changes in laboratory parameters after index treatment (V3) and as a function of time will be analysed and compared between randomization arms.
Laboratory parameter (ALT) | through study completion, an average of 1 year
  Changes in laboratory parameters after index treatment (V3) and as a function of time will be analysed and compared between randomization arms.
Laboratory parameter (GGT) | through study completion, an average of 1 year
  Changes in laboratory parameters after index treatment (V3) and as a function of time will be analysed and compared between randomization arms.
Pruritus as reported by patients on a scale from 0 ("no itching") to 10 ("worst imaginable itching"). | through study completion, an average of 1 year
  Pruritus will be analysed as a function of time.

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Hoffmeister, Prof.Dr.med., Principal Investigator — Universitätsklinikum Leipzig; Bereich Gastroenterologie
Locations (20):
- Germany (20):
  - Uniklinik RWTH Aachen, Medizinische Klinik III, Aachen
  - Universitätsklinikum Augsburg; III. Med. Klinik, Augsburg
  - Vivantes Netzwerk für Gesundheit GmbH, Klinikum Friedrichshain, Innere Medizin/Gastroenterologie, Berlin
  - Universitatsklinikum Bonn, Medizinische Klinik und Poliklinik I, Bonn
  - Universitätsklinikum Frankfurt, Medizinische Klinik 1, Frankfurt
  - Universitätsklinikum Freiburg, Medizinische Klinik II, Abteilung Gastroenterologie, Hepatologie, Endokrinologie & lnfektiologie, Freiburg im Breisgau
  - Universitätsmedizin Greifswald Klinik für Innere Medizin A, Greifswald
  - Site: Martin-Luther-Universitat Halle-Wittenberg, Universitätsklinik und Poliklinik für Innere Medizin I, Halle
  - Klinikum Hanau; Klinik für Gastroenterologie, Diabetologie und Infektiologie, Hanau
  - KRH Klinikum Siloah, Klinik für Gastroenterologie, Hanover
  - Klinikum St. Georg gGmbH; Klinik für Gastroenterologie, Hepatologie, Diabetologie und Endokrinologie, Leipzig
  - University Hospital of Leipzig, Department of Gastroenterology, Leipzig
  - RKH Kliniken Ludwigsburg- Bietigheim gGmbH, Klinik für Innere Medizin, Gastroenterologie, Hämato-Onkologie, Diabetologie und Infektiologie, Ludwigsburg
  - Universitätsmedizin Mannheim, II. Medizinische Klinik, Mannheim
  - Universitätsklinikum Gießen und Marburg GmbH (UKGM); Klinik für Innere Medizin mit den Schwerpunkten Gastroenterologie, Endokrinologie, Stoffwechsel und klinische Infektiologie, Marburg
  - Klinikum der LMU München, Medizinische Klinik II, Campus Großhadern, München
  - Universitlitsklinikum Munster Medizinische Klinik B (Gastroenterologie, Hepatologie, Endokrinologie, Klinische lnfektiologie), Münster
  - Klinikum Nürnberg Nord; Gastroenterologie/ Endokrinologie, Nuremberg
  - Robert-Bosch-Krankenhaus (RBK) Stuttgart; Gastroenterologie, Hepatologie und Endokrinologie, Stuttgart
  - Universitätsklinikum Tübingen, Medizinische Klinik I, Tübingen

IPD SHARING:
Plan to Share IPD: No